CLINICAL TRIAL: NCT02621177
Title: A Multi-center, Randomized, Double-blind Phase III Clinical Trial to Assess the Immunogenicity and Safety of 'NBP607(Trivalent Inactivated Cell Culture-derived Influenza Vaccine)' in Healthy Children and Adolescents Aged 6 Month ~ 18 Years)
Brief Title: Study of Egg-derived Influenza Vaccine and Cell Culture-derived Influenza Vaccine in Healthy Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP607_FluC_III_2013
Record Dates: First submitted 2015-11-30; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBP607 (Experimental): Trivalent Inactivated Cell Culture-derived Influenza Vaccine
  Interventions: Biological: NBP607
- Agrippal S1 (Active Comparator): Trivalent Inactivated Egg-derived Influenza Vaccine
  Interventions: Biological: Agrippal S1

INTERVENTIONS:
Biological: NBP607 — For subjects 6 months to 8 years of age, single intramuscular dose for primed subjects, two doses for unprimed subjects. For subjects 9 to 18 years of age, single intramuscular dose (0.25mL/0.5 mL)
  Arms: NBP607
Biological: Agrippal S1 — For subjects 6 months to 8 years of age, single intramuscular dose for primed subjects, two doses for unprimed subjects. For subjects 9 to 18 years of age, single intramuscular dose (0.25mL/0.5 mL)
  Arms: Agrippal S1

SUMMARY:
This study is a multi-center, randomized, double-blind Phase III clinical trial. The aim of the study is to describe the immunogenicity and safety of the trivalent cell culture-derived influenza vaccine compared to the trivalent egg-derived influenza vaccine among subjects.

DETAILED DESCRIPTION:
Subjects are randomly assigned in a 4:1 ratio to NBP607-QIV versus Agrippal S1. To assess the immunogenicity, antibody levels are evaluated by hemagglutination inhibition(HI) assay from sera obtained at pre-vaccination and 28 days post-vaccination. To assess the safety, solicited adverse events for 7 days post-vaccination and unsolicited adverse events for 28 days post-vaccination are assessed and reported. The serious adverse events are collected during 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and adolescents aged 6 months to 18 years.
* Those who was born after normal pregnancy period(37 weeks) for aged 6 months to 2 years.
* Those whose legally acceptable representative have given written consent to participate in the study and comply with all study requirements.

Exclusion Criteria:

* Subjects who are hypersensitive to any component of vaccine, i.e., eggs, chicken or chicken products.
* Subjects with immune deficiency disorder.
* History of Guillain-Barre syndrome.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Subjects who experienced fever within 72 hours before vaccination or with the febrile disease(exceeding 38.0℃) on screening day or with any acute respiratory infection.
* Subjects who had received immunosuppressant or immune-modifying drug within 3 months before screening.
* Subjects who had received blood products or immunoglobulin within 3 months before screening.
* Subjects who had received influenza vaccination within 6 months prior to the screening.
* Subjects who had received other vaccination within a month before screening, or those who had another vaccination scheduled within a month after study vaccination.
* Subjects who had participated in other clinical trial within 4 weeks prior to study vaccination.
* Subjects who had done blood donation within a week prior to study vaccination or planned blood donation within 7 months after study vaccination.
* Subjects with clinically significant chronic disease or malignant cancer.
* Pregnant women, breast-feeding women.
* Any other condition which, in the opinion of the Investigator, prevents the subject from participating in the study.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 385 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
CHMP criteria | At Day 28 post-vaccination
  Seroprotection rate > 70%, Seroconversion rate > 40%, GMR > 2.5

SECONDARY OUTCOMES:
Immunogenicity in subjects with a pre-vaccination HI antibody titer < 1:80 | At Day 28 post-vaccination
Immunogenicity compared to control group | At Day 28 post-vaccination
Incidence rate of Advers Event (AE) | During 7 days post-vaccination for Solicited AE and during 28 days post-vaccination for Unsolicited AE
  Including Solicited Local AE, Solicited Systemic AE, and Unsolicited AE
Incidence rate of Severe Adverse Event (SAE) | During 6 months post-vaccination
Vital Sign | At Day 0 and at Day 28 post-vaccination
Physical Examination | At Day 0 and at Day 28 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kyung Kim, Study Chair — Korea University Ansan Hospital; Ui Yoon Choi, Principal Investigator — Catholic University of Korea Saint Paul's Hospital; Chi Eun Oh, Principal Investigator — Kosin University Gospel Hospital; Byung Wook Eun, Principal Investigator — Eulji General Hospital; Taek Jin Lee, Principal Investigator — CHA University; Ki Hwan Kim, Principal Investigator — Severance Children's Hospital; Dong Ho Kim, Principal Investigator — Korea Institute of Radiological and Medical Science; Nam Hee Kim, Principal Investigator — Inje University Ilsan Paik Hospital; Dae Sun Jo, Principal Investigator — Chonbuk National University Hospital; Seon Hee Shin, Principal Investigator — Hallym University Dongtan Sacred Heart Hospital